CLINICAL TRIAL: NCT03167684
Title: The Effect of Oral Appliance Therapy on Cardiometabolic Outcomes in Patients With Type 2 Diabetes and Obstructive Sleep Apnea: A Pilot RCT
Brief Title: Effect of Oral Appliance Therapy on Glucose Levels in Patients With T2DM and OSA: A Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Sushmita Pamidi, Clinician Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-2769
Record Dates: First submitted 2017-05-21; First posted 2017-05-30 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Sleep Apnea, Obstructive; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2 | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral appliance therapy (Experimental): Oral appliance (SomnoMed) worn nightly
  Interventions: Device: Oral appliance therapy
- Control (No Intervention): Sham oral appliance device

INTERVENTIONS:
Device: Oral appliance therapy — Fitted oral appliance
  Other Names: Mandibular advancement device
  Arms: Oral appliance therapy

SUMMARY:
This study will evaluate the impact on blood glucose of the use of an oral appliance to treat obstructive sleep apnea (OSA) in individuals with Type 2 diabetes. An oral appliance is similar to a sports mouth guard or an orthodontic retainer and is an alternative treatment to continuous positive airway pressure (CPAP) for OSA. Oral appliance therapy has not been evaluated in patients with Type 2 diabetes with respect to glycemic outcomes. This will be a 1:1 randomized controlled trial: The experimental group will receive the oral appliance and the control group will receive a sham device over the course of approximately 5 months.

DETAILED DESCRIPTION:
OSA is quite common in individuals with T2DM, occurring in as many as 60-80% of patients. The standard treatment for OSA is with the use of a CPAP machine. The CPAP provides an air pressure to keep the airways opened during sleep so that a person with OSA can breathe normally. When used appropriately, the CPAP improves sleepiness and quality of life. However, about half of the patients who receive a CPAP prescription cannot tolerate it and thus remain untreated and are potentially at increased cardiovascular and diabetes risk. In light of this, this study aims to see if the use of an alternative treatment for OSA, oral appliance therapy, where adherence is generally superior to CPAP, will improve cardiometabolic outcomes in individuals with Type 2 diabetes. This pilot trial will primarily examine feasibility and assess recruitment rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM using current Canadian guidelines
* OSA with AHI > 10 events/hour using current American Academy of Sleep Medicine (AASM) criteria for scoring respiratory events

Exclusion Criteria:

* On treatment for OSA within the past 3 months
* Professional drivers or patients with an increased risk of driving-related accidents from clinical interview or severe subjective sleepiness (Epworth sleepiness scale greater than 15)
* Sleep apnea with any of the following features: highly severe OSA (AHI>50 and oxygen desaturation index > 50), severe hypoxemia (SpO2<80% for >10% of recording time), central sleep apnea or Cheyne-Stokes respirations with a central apnea index >10 events/hour
* Coexisting sleep disorder other than OSA
* Active cardiovascular disease, including angina, arrhythmia or congestive heart failure
* Insufficient dentition or significant periodontal disease or other contraindication for OAT as determined by dentist qualified in OSA treatment
* Active and significant psychiatric disease
* BMI>35
* Regular use of sedatives or narcotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rates | End of study (Week 20)
  feasibility of study in T2DM
Glycemic control (mean 24-hour and nocturnal glucose) | End of study (week 20)
  24-hour continuous glucose monitoring

SECONDARY OUTCOMES:
Blood pressure | End of study (Week 20)
  Measurement of clinic blood pressure
Glucose variability | End of study (Week 20)
  Continuous glucose monitoring system (ipro2, Medtronic)
Changes in insulin or diabetes medication doses | End of study (Week 20)
  Reporting of dose change by participant or treating physician.
Systemic inflammation | End of study (Week 20)
  hs-CRP

OTHER OUTCOMES:
Oral appliance therapy adherence | Monitored from Week 0 to week 20 (8 week titration + 12 week treatment)
  Measured by a chip embedded in the oral appliance
Subjective sleep quality | Screening or baseline (Week -4), Week 12 and End of study (Week 20)
  Sleep questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sushmita Pamidi, MD MSc, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- McGill University Health Centre - Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Towards meta-analysis data